CLINICAL TRIAL: NCT04321174
Title: COVID-19 Ring-based Prevention Trial With Lopinavir/Ritonavir
Acronym: CORIPREV-LR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CORIPREV-1
Record Dates: First submitted 2020-03-18; First posted 2020-03-25 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Infections; Post-exposure Prophylaxis
MeSH Terms: conditions — Coronavirus Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lopinavir/ritonavir (Experimental): This arm will receive oral lopinavir/ritonavir 400/100 mg (or equivalent weight-based dosing) twice daily for 14 days.
  Interventions: Drug: Lopinavir/ritonavir
- Control (No Intervention): This arm will receive no intervention.

INTERVENTIONS:
Drug: Lopinavir/ritonavir — The intervention is a 14-day course of LPV/r 400/100 mg orally twice daily, or equivalent weight-based dosing, to be initiated as soon as possible (within 1-7 days) after the last exposure.
  Other Names: Kaletra; Aluvia
  Arms: Lopinavir/ritonavir

SUMMARY:
COVID-19 has rapidly evolved into a generalized global pandemic. Post-exposure prophylaxis (PEP) against on COVID-19 was identified as an urgent research priority by the WHO, and lopinavir/ritonavir (LPV/r) is a promising candidate for both COVID-19 treatment and PEP, with a good safety profile and global availability. This is a cluster randomized controlled trial (RCT) of oral LPV/r as PEP against COVID-19, that will address the immediate need for preventive interventions, generate key data on COVID-19 transmission, and serve as a research platform for future vaccines and preventive agents.

ELIGIBILITY:
Inclusion Criteria:

1. High risk close contact with a confirmed COVID-19 case during their symptomatic period, including one day before symptom onset, within the past 1-7 days. High risk close contact is defined as any of the following exposures without the consistent appropriate use of recommended personal protective equipment:

   1. Provided direct care for the index case
   2. Had close physical contact with the index case
   3. Lived with the index case
   4. Had close contact (within 2 metres), without direct physical contact, for a prolonged period of time
   5. Had direct contact with infectious body fluids, including oral secretions, respiratory secretions, or stool.
2. Successfully contacted by the study team within 24 hours of study team notification of the relevant index COVID-19 case. This time window is necessary because the efficacy of PEP may be dependent on the timing of its initiation, and because randomization of a ring cannot be delayed while awaiting response from contacts that cannot be rapidly reached.
3. Age ≥6 months, since the safety and pharmacokinetic profiles of LPV/r in pediatric patients below the age of 6 months have not been established.
4. Ability to communicate with study staff in English

Exclusion Criteria:

1. Known hypersensitivity/allergy to lopinavir or ritonavir.
2. Current use of LPV/r for the treatment or prevention of HIV infection.
3. Receipt of LPV/r in the context of this trial or any other trial of COVID-19 PEP within 2 days or less prior to the last known contact with the index COVID-19 case. The two day time window is intended to ensure that exposure would not have occurred in the presence of clinically relevant drug levels (five times the elimination half-life of LPV/r, which is estimated at 4-6 hours with prolonged use).
4. Baseline respiratory tract specimen positive for COVID-19. Randomized participants whose baseline samples subsequently show COVID-19 will have study drug discontinued but still remain under observation.
5. Current breastfeeding, due to potential for serious adverse reactions in nursing infants exposed to LPV/r
6. Concomitant medications with prohibited drug interactions with LPV/r that cannot be temporarily suspended/replaced, including but not restricted to: 37

   * alfuzosin (e.g. Xatral®)
   * amiodarone (e.g. Cordarone™)
   * apalutamide (e.g. Erleada™)
   * astemizole*, terfenadine*
   * cisapride*
   * colchicine, when used in patients with renal and/or hepatic impairment
   * dronedarone (e.g., Multaq®)
   * elbasvir/grazoprevir (e.g., ZepatierTM)
   * ergotamine* (e.g. Cafergot®*), dihydroergotamine (e.g. Migranal®), ergonovine, methylergonovine*
   * fusidic acid (e.g., Fucidin®), systemic*
   * lurasidone (e.g., Latuda®), pimozide (e.g., Orap®*)
   * neratinib (e.g., Nerlynx®)
   * sildenafil (e.g., Revatio®)
   * triazolam (e.g. Halcion®), midazolam oral*
   * rifampin (e.g. Rimactane®*, Rifadin®, Rifater®*, Rifamate®*)
   * St. John's Wort
   * Tadalafil (e.g. Adcirca®)
   * venetoclax (e.g. Venclexta®)
   * lovastatin (e.g., Mevacor®*), lomitapide (e.g., JuxtapidTM) or simvastatin (e.g., Zocor®)
   * vardenafil (e.g., Levitra® or Staxyn®)
   * salmeterol (e.g., Advair® or Serevent®)

     * denotes products not marketed in Canada

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Microbiologic evidence of infection | 14 days
  The primary outcome is microbiologically confirmed COVID-19 infection, ie. detection of viral RNA in a respiratory specimen (mid-turbinate swab, nasopharyngeal swab, sputum specimen, saliva specimen, oral swab, endotracheal aspirate, bronchoalveolar lavage specimen) by day 14 of the study.

SECONDARY OUTCOMES:
Adverse events | 90 days
  a) Adverse events: as defined using the DAIDS Table for Grading the Severity of Adverse Events, at 7, 14, 28 & 90 days
Symptomatic COVID-19 disease | 14 days
  fever, cough or other respiratory/ systemic symptoms (including but not limited to fatigue, myalgias, arthralgias, shortness of breath, sore throat, headache, chills, coryza, nausea, vomiting, diarrhea) by day 14 in a patient with laboratory confirmed infection, combined with microbiologic confirmation of COVID-19 infection in the participant.
Seropositivity | 28 days
  Reactive serology to SARS-CoV-2
Days of hospitalization attributable to COVID-19 disease | 90 days
  The number of days (or partial days) spent admitted to an acute care hospital will be tabulated both at day 28 and day 90
Respiratory failure requiring ventilatory support attributable to COVID-19 disease | 90 days
  The number of days (or partial days) requiring i) non-invasive and ii) endotracheal intubation with ventilation will be tabulated both at day 28 and day 90.
Mortality | 90 days
  Death attributable to COVID-19 disease and all-cause mortality
Short-term psychological impact of exposure to COVID-19 disease | 28 days
  Short-term psychological distress will be measured using the K10, with a standard cutoff score of ≥16.
Long-term psychological impact of exposure to COVID-19 disease | 90 days
  Long-term impact will be measured at day 90 using the Impact of Event Scale, a validated measure of traumatic stress response, using a standard cutoff score of ≥26
Health-related quality of life | 90 days
  Health-related quality of life will be measured using the EQ-5D-5L (EuroQol-5D). The EQ-5D consists of two pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The tool will be administered to participants at 1, 14, 28 and 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Tan, MD FRCPC PhD, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
TBA

REFERENCES:
- [Derived] Tan DHS, Chan AK, Juni P, Tomlinson G, Daneman N, Walmsley S, Muller M, Fowler R, Murthy S, Press N, Cooper C, Lee T, Mazzulli T, McGeer A. Post-exposure prophylaxis against SARS-CoV-2 in close contacts of confirmed COVID-19 cases (CORIPREV): study protocol for a cluster-randomized trial. Trials. 2021 Mar 22;22(1):224. doi: 10.1186/s13063-021-05134-7. PMID 33752741
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583
- [Derived] Sultana J, Crisafulli S, Gabbay F, Lynn E, Shakir S, Trifiro G. Challenges for Drug Repurposing in the COVID-19 Pandemic Era. Front Pharmacol. 2020 Nov 6;11:588654. doi: 10.3389/fphar.2020.588654. eCollection 2020. PMID 33240091